CLINICAL TRIAL: NCT01248754
Title: A Phase II Study Using 18F-FDOPA Positron Emission Tomography Imaging for Neurosurgery and Assessment of Surgical Resection
Brief Title: Positron Emission Tomography (PET) With 3,4-dihydroxy-6-18F-fluoro-L-enylalanine (18F-FDOPA) Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alan Nichol (Other)
Responsible Party: Sponsor-Investigator, Alan Nichol, Radiation Oncologist, British Columbia Cancer Agency
Organization: British Columbia Cancer Agency (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H10-02888
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Cancer (High-grace Glioma)
Keywords: Neurosurgery; Neuronavigation; Positron emission tomography; FDOPA
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 18F-DOPA PET imaging (Experimental): Subjects will undergo preoperative 18F-FDOPA PET imaging, which will be used in neuronavigation software to guide resection of their high-grade glioma. Postoperative 18F-FDOPA PET imaging will be obtained to determine the extent of resection.
  Interventions: Procedure: Surgical neuronavigation with 18F-DOPA PET imaging

INTERVENTIONS:
Procedure: Surgical neuronavigation with 18F-DOPA PET imaging — Subjects will undergo preoperative 18F-FDOPA PET imaging, which will be used in neuronavigation software to guide resection of their high-grade glioma. Postoperative 18F-FDOPA PET imaging will be obtained to determine the extent of resection.

SUMMARY:
The 18F-FDOPA PET tracer is an amino acid analogue that can be used to visualize high-grade glioma not clearly identified on diagnostic MRI. Use of 18F-FDOPA PET will permit neurosurgeons to achieve a complete resection more frequently.

ELIGIBILITY:
Inclusion Criteria:

* Contrast-enhancing mass on diagnostic brain CT or MRI strongly suggesting a diagnosis of WHO grade III or IV glioma
* Karnofsky Performance status (KPS) ≥ 70
* Age ≥18 years
* Subject is able to understand and consent to study
* Glomerular filtration rate (GFR) ≥ 45 ml/minute

Exclusion Criteria:

* Indication for urgent craniotomy to relieve mass effect
* Only stereotactic biopsy indicated because tumour is located in eloquent brain.
* The enhancement on the T1 MRI sequence involves or abuts the basal ganglia
* Previous intracranial malignancy or any invasive malignancy unless free of disease > 5 years
* Prior cranial irradiation
* Contra-indications to systemic radiation exposure: pregnancy or breast feeding
* Subject exceeds the weight limit of the PET scanner bed (204.5 kg)
* Subjects taking medication such as Levodopa for the treatment of Parkinson's Disease
* Allergies or other contraindication to CT contrast or MRI contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects that have a complete resection of the volume of 18F-FDOPA PET tracer on their postoperative 18F-FDOPA PET scan. | Less than 72 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Alan Nichol, MD, Principal Investigator — British Columbia Cancer Agency
Locations (3):
- Canada (3):
  - Lions Gate Hospital, North Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - BC Cancer Agency, Vancouver, British Columbia

REFERENCES:
- See also: BC Cancer Agency — http://www.bccancer.bc.ca
- See also: UBC Department of Surgery — http://www.surgery.ubc.ca/